CLINICAL TRIAL: NCT00907699
Title: Study of Epithelial Growth Factor Receptor Mutations in Tumor Specimens and Blood Samples From Patients With Non-Small Cell Lung Cancer Enrolled on Clinical Trial CASE-2507
Brief Title: Laboratory Study Using Samples From Patients With Non-Small Cell Lung Cancer Treated on Clinical Trial CASE-2507
Status: Withdrawn | Type: Observational
Why Stopped: Slow Accrual
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CASE9507; P30CA043703 (NIH); CASE9507 (Other: Case Comprehensive Cancer Center)
Record Dates: First submitted 2009-05-21; First posted 2009-05-22 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — In Situ Hybridization, Fluorescence; Gene Expression Profiling; Polymerase Chain Reaction; Reverse Transcriptase Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — This laboratory study is looking at biomarkers in tumor tissue and blood samples from patients with non-small cell lung cancer.
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Genetic: DNA analysis — DNA is extracted from tumor samples. Genomic DNA is analyzed using real-time PCR/ reverse transcriptase PCR analysis and/or FISH analysis in order to study resistance mechanisms such as secondary EGFR mutations and the c-MET and PI3K pathways.
Genetic: RNA analysis — RNA is extracted from tumor samples. RNA is analyzed using TaqMan quantitative PCR in order to determine the copy number of EGFR expressed in these tissues. Peripheral blood samples are used to isolate peripheral blood mononuclear cells positive for epithelial cell adhesion molecule (EpCAM).
Genetic: fluorescence in situ hybridization — DNA and RNA are extracted from tumor samples. Genomic DNA is analyzed using real-time PCR/ reverse transcriptase PCR analysis and/or FISH analysis in order to study resistance mechanisms such as secondary EGFR mutations and the c-MET and PI3K pathways. RNA is analyzed using TaqMan quantitative PCR in order to determine the copy number of EGFR expressed in these tissues. Peripheral blood samples are used to isolate peripheral blood mononuclear cells positive for epithelial cell adhesion molecule (EpCAM).
Genetic: gene expression analysis — DNA and RNA are extracted from tumor samples. Genomic DNA is analyzed using real-time PCR/ reverse transcriptase PCR analysis and/or FISH analysis in order to study resistance mechanisms such as secondary EGFR mutations and the c-MET and PI3K pathways. RNA is analyzed using TaqMan quantitative PCR in order to determine the copy number of EGFR expressed in these tissues. Peripheral blood samples are used to isolate peripheral blood mononuclear cells positive for epithelial cell adhesion molecule (EpCAM).
Genetic: mutation analysis — DNA and RNA are extracted from tumor samples. Genomic DNA is analyzed using real-time PCR/ reverse transcriptase PCR analysis and/or FISH analysis in order to study resistance mechanisms such as secondary EGFR mutations and the c-MET and PI3K pathways. RNA is analyzed using TaqMan quantitative PCR in order to determine the copy number of EGFR expressed in these tissues. Peripheral blood samples are used to isolate peripheral blood mononuclear cells positive for epithelial cell adhesion molecule (EpCAM).
Genetic: polymerase chain reaction — DNA and RNA are extracted from tumor samples. Genomic DNA is analyzed using real-time PCR/ reverse transcriptase PCR analysis and/or FISH analysis in order to study resistance mechanisms such as secondary EGFR mutations and the c-MET and PI3K pathways. RNA is analyzed using TaqMan quantitative PCR in order to determine the copy number of EGFR expressed in these tissues. Peripheral blood samples are used to isolate peripheral blood mononuclear cells positive for epithelial cell adhesion molecule (EpCAM).
Genetic: reverse transcriptase-polymerase chain reaction — DNA and RNA are extracted from tumor samples. Genomic DNA is analyzed using real-time PCR/ reverse transcriptase PCR analysis and/or FISH analysis in order to study resistance mechanisms such as secondary EGFR mutations and the c-MET and PI3K pathways. RNA is analyzed using TaqMan quantitative PCR in order to determine the copy number of EGFR expressed in these tissues. Peripheral blood samples are used to isolate peripheral blood mononuclear cells positive for epithelial cell adhesion molecule (EpCAM).
Other: laboratory biomarker analysis — DNA and RNA are extracted from tumor samples. Genomic DNA is analyzed using real-time PCR/ reverse transcriptase PCR analysis and/or FISH analysis in order to study resistance mechanisms such as secondary EGFR mutations and the c-MET and PI3K pathways. RNA is analyzed using TaqMan quantitative PCR in order to determine the copy number of EGFR expressed in these tissues. Peripheral blood samples are used to isolate peripheral blood mononuclear cells positive for epithelial cell adhesion molecule (EpCAM).

SUMMARY:
RATIONALE: Studying samples of blood and tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and RNA and identify biomarkers related to cancer.

PURPOSE: This laboratory study is looking at biomarkers in tumor tissue and blood samples from patients with non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Identify mutations in epidermal growth factor receptor (EGFR) in non-small cell lung cancer specimens from clinical trial CASE-2507.
* Investigate EGFR DNA copy-number changes.
* Determine abnormalities of other pathways, such as the c-MET and PI3K pathways as potential mechanisms of resistance.

OUTLINE: This is a multicenter study.

DNA and RNA are extracted from tumor samples. Genomic DNA is analyzed using real-time PCR/ reverse transcriptase PCR analysis and/or FISH analysis in order to study resistance mechanisms such as secondary EGFR mutations and the c-MET and PI3K pathways. RNA is analyzed using TaqMan quantitative PCR in order to determine the copy number of EGFR expressed in these tissues. Peripheral blood samples are used to isolate peripheral blood mononuclear cells positive for epithelial cell adhesion molecule (EpCAM).

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Eligible for and concurrently enrolled on clinical trial CASE-2507

PATIENT CHARACTERISTICS:

* Willing and able to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures
* Normal coagulation profile and platelet count > 100,000/mm³*
* Not pregnant NOTE: *For patients who have not had a second biopsy procedure already at the time of progression on erlotinib hydrochloride therapy and require a research biopsy.

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No concurrent anticoagulants (e.g., warfarin or low-molecular weight heparin)
* No concurrent antiplatelet therapy (e.g., aspirin, clopidogrel, or other antiplatelet agents)* NOTE: *For patients who have not had a second biopsy procedure already at the time of progression on erlotinib hydrochloride therapy and require a research biopsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-08; Primary Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Predictive value of T790M mutation status of the second biopsy (before maintenance therapy on CASE-2507) on progression-free survival (PFS) | At the time of the second biopsy or surgical procedures
Difference of PFS between those with and without T790M mutation | At the time of the second biopsy or surgical procedures
Difference of clinical response rate between T790M mutation statuses | At the time of the second biopsy or surgical procedures
Predictive value of mutation status on clinical response | At the time of the second biopsy or surgical procedures
Association between T790M mutation and baseline clinical-pathological factors and smoking status | At the time of the second biopsy or surgical procedures

CONTACTS AND LOCATIONS:
Overall Officials: Afshin Dowlati, MD, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center